CLINICAL TRIAL: NCT02370082
Title: A Prospective, Single-Arm, Multi-Site, Clinical Evaluation of the SAVI SCOUT® Surgical Guidance System for the Location of Non-Palpable Breast Lesions During Excision
Brief Title: SAVI SCOUT Clinical Evaluation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cianna Medical, Inc. (Industry)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019820
Record Dates: First submitted 2015-02-02; First posted 2015-02-24 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-02

CONDITIONS: Breast Neoplasm
Keywords: lumpectomy; breast conserving surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAVI SCOUT device (Experimental): SAVI SCOUT device used to localize breast lesion which will then be removed surgically. The SAVI SCOUT is the intervention for localization of breast lesions.
  Interventions: Device: Localization of breast lesion

INTERVENTIONS:
Device: Localization of breast lesion — localization of breast lesion for removal

SUMMARY:
The purpose of this study is to evaluate the performance of the SAVI SCOUT® Surgical Guidance System (SAVI SCOUT). The SAVI SCOUT is a medical device, used to provide real-time guidance during localized excisional biopsy or lumpectomy procedures, by helping the surgeon locate and remove the desired tissue (i.e., the lesion and surrounding normal tissue). The SAVI SCOUT has been 510K cleared.

The SAVI SCOUT is intended to assist surgeons in the location and retrieval of a non-palpable abnormality as localized by radiographic or ultrasound methods. In this study, the ability of the SAVI SCOUT to guide surgeons to find a lesion will be evaluated instead of the standard technique of wire localization.

DETAILED DESCRIPTION:
Using radiography or ultrasound guidance, the SAVI SCOUT reflector will be placed percutaneously up to 7 days prior to the scheduled excisional procedure. During surgical excision, the SAVI SCOUT system will be used to locate the reflector, which will be removed along with the surrounding breast tissue.

Final data analysis will be completed within 1 month after the last patient is treated.

Final assessment of the surgical results will be completed by the surgeon during a routine follow-up visit within 1 month following the surgical excision or lumpectomy procedure.

Main Objective: to show that the SAVI SCOUT technique can be used to safely and effectively locate a non-palpable breast lesion during a localized excisional biopsy or lumpectomy procedure.

Up to 10 sites and 150 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* • Patient has a non-palpable breast lesion that requires excision

  * Lesion depth ≤ 3 cm from the skin surface in the supine position
  * Patient is scheduled for excision or BCT at a participating institution
  * Patient is between the ages of 18 and 90 years
  * Patient is female
  * Patient is willing and able to comply with all study procedures and be available to follow-up for the duration of the study
  * For lesions requiring multiple reflectors for localization, they must allow for reflectors to be placed ≥ 1cm from one another relative to the coronal plane Subject Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

* Patient had a previous ipsilateral breast cancer
* Patient has multicentric breast cancer
* Patient has Stage IV breast cancer
* Patient has been treated with neoadjuvant chemotherapy
* Patient is pregnant or lactating

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Success rate of reflector placement | intraoperative
  How often the reflector can be successfully placed

SECONDARY OUTCOMES:
Amount of tissue excised | Will be assessed by pathologist during standard pathology assessment which occurs 24-48 hours after surgery
  Pathologic assessment of how much tissue was removed
Percent of cases with clear margins • Percent of cases requiring a second operation | Upon completion of pathologic assessment-which will occur within 24-48 hours after surgery
  How often patients are not required to have repeat procedures

CONTACTS AND LOCATIONS:
Overall Officials: Charles Cox, MD, Principal Investigator — University of South Florida